

# Clinical, Radiographic and Patient-reported Outcomes Associated with the Use of the Navio<sup>o</sup> Robotic-assisted Surgical System in Total Knee Arthroplasty

Protocol Number: 17-NPFS-04

Protocol Date: 19SEP2017

Protocol Version: Version 2.0

Study Product Name: Navio \* Robotic-assisted Surgical System

Sponsor: Smith & Nephew, Inc.

1450 E. Brooks Road Memphis, TN 38116

US

#### **Nondisclosure Statement**

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith & Nephew and its manufacturers. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any mean without prior written permission from Smith & Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith & Nephew.



#### Table of Contents

| ABBR | eviations & Definitions | 5 |
|-------|-------------------------------------------|----|
| Proto | ocol Synopsis: | 6 |
| 1. | BACKGROUND AND STUDY RATIONALE | 8 |
| 1.1. | Background | 8 |
| 1.2. | Study Rationale | 8 |
| 2. | STUDY OBJECTIVES. | 8 |
| 2.1. | Primary Objective | 8 |
| 2.2. | Secondary Objectives | 8 |
| 3. | STUDY ENDPOINTS | 8 |
| 3.1. | Primary Endpoint | 8 |
| 3.2. | Secondary Endpoints | 9 |
| 3.3. | Safety Endpoints | 9 |
| 5.1. | Surgical Technique | 11 |
| 6. | STUDY POPULATION | 11 |
| 6.1. | Subject Screening & Enrollment | 11 |
| 6.2. | Subject Inclusion Criteria | 11 |
| 6.3. | Subject Exclusion Criteria | 12 |
| 7. | STUDY PROCEDURES. | 13 |
| 7.1. | Study Schematic | 13 |
| 7.2. | Pre-Operative Visit | 13 |
| 7.3. | Surgery | 13 |
| 7.4. | One Month Post-Operative Visit | 14 |
| 8. | SUBJECT COMPLETION AND DISPOSITION | 14 |
| 8.1. | Screening | 14 |
| 8.2. | Enrolled Subject | 14 |
| 8.3. | Conditions for Study Termination | 14 |
| Α. | Screening Failure | 14 |
| B. | Voluntary Withdrawal | 14 |
| C. | Lost to Follow-Up | 15 |
| D. | Study Termination by Investigator/Sponsor | 15 |
| E. | Pregnancy | 15 |
| F. | Study Site Discontinuation | 15 |
| 9. | SAFETY REPORTING | 15 |



| 9.1. | Definitions for safety reporting | 15 |
|-------|-----------------------------------------------------|----|
| A. | Adverse Event (AE) | 16 |
| B. | Serious Adverse Event (SAE) | 16 |
| C. | Adverse Device Effect (ADE) | 16 |
| D. | Serious Adverse Device Effect (SADE) | 16 |
| E. | Unanticipated Serious Adverse Device Effect (USADE) | 16 |
| F. | Device Deficiency | 16 |
| G. | Revisions | 17 |
| 9.2. | Safety: Investigator's Responsibilities | 17 |
| 9.3. | Timelines for Submission of Safety Information: | 17 |
| 9.4. | Safety reporting: Sponsor's Responsibilities | 18 |
| 10. | STATISTICAL PROCEDURES | 18 |
| 10.1. | Sample size calculation | 18 |
| 10.2. | . General Statistical Considerations | 18 |
| 10.3. | . Missing Data | 19 |
| 10.4. | . Analysis Populations | 19 |
| 10.5. | . Analysis of Primary Endpoint | 19 |
| 10.6. | . Analysis of Secondary Endpoints: | 19 |
| 10.7. | Analysis of Safety Endpoints: | 20 |
| 11. | ETHICAL CONSIDERATIONS | 20 |
| 11.1. | Ethical Approval | 20 |
| 11.2. | Protocol Amendments | 20 |
| 11.3. | Informed Consent | 20 |
| 11.4. | Risk – Benefit Analysis | 20 |
| Α. | Study Related Risks | 20 |
| B. | Study Related Benefits | 21 |
| 12. | MONITORING PROCEDURES | 21 |
| 12.1. | Source Documentation | 21 |
| 12.2. | . Direct Access | 21 |
| 12.3. | . Site Qualification Visit | 21 |
| 12.4. | . Site Initiation Visit | 21 |
| 12.5. | . Interim Monitoring Visits | 22 |
| 12.6. | . Closeout Visit | 22 |
| 12.7. | . Sponsor Audits and Regulatory Inspection | 22 |
| 12.8. | . Data Handling and Record Keeping Requirements | 22 |



| 12.9 | Data Recording and Record Retention | .22 |
|-------|-------------------------------------------|-----|
| 13. | DEVIATIONS FROM PROTOCOL | .23 |
| 13.1. | Protocol Deviation Reporting Requirements | .23 |
| 14. | Publication policy | .23 |
| Bibli | OGRAPHY | .24 |
| | endix 1 | |
| JOU | RNEY II BCS and CR Component Part Numbers | .28 |



#### ABBREVIATIONS & DEFINITIONS

| AE | Adverse Event |
|---|---|
| ADE | Adverse Device Effect |
| AP | Anteroposterior |
| CAPA | Corrective and Preventive Action |
| CRO Contract Research Organization | |
| CRF | Case Report Form |
| EC | Ethics Committee |
| EQ-5D | EuroQuol 5D |
| FDA | Food and Drug Administration |
| FU | Follow-Up |
| GCP | Good Clinical Practice |
| ICF | Informed Consent Form |
| | International Conference on Harmonisation of Technical Requirements for Registration of |
| ICH | Pharmaceuticals for Human Use |
| IRB | Institutional Review Board |
| ITT | Intention to Treat Population |
| KSS | Knee Society Score |
| PI | Principal Investigator |
| PP | Per-protocol Population |
| QoL | Quality of life |
| SAE | Serious Adverse Event |
| SADE | Serious Adverse Device Effect |
| TKA | Total Knee Arthroplasty |
| USADE | Unanticipated Serious Adverse Device Effect |



## **Protocol Synopsis:**

| Title of Study: | Clinical, Radiographic, and Patient-reported Outcomes associated with the use of the Navio° Robotic-assisted Surgical System in Total Knee Arthroplasty |
|---|---|
| Study Type: | Evidence Generation |
| Study Device: | Navio <sup>o</sup> Robotic-assisted Surgical System |
| Study Purpose: | To demonstrate superior accuracy with the Navio° Robotic-assisted Surgical System in achieving desired post-operative mechanical alignment, compared to TKA procedures using standard instruments, as well as to document clinical and patient-reported outcomes in subjects receiving TKA with the Navio° system. |
| Study Design: | Multicenter, prospective single-arm cohort study with historical control. |
| Primary Endpoint: | Post-operative Mechanical Alignment (percentage of subjects achieving target alignment, defined as $\pm 3^{\circ}$ from target) at one month post-operative. |
| Secondary<br>Endpoints: | <ul> <li>Implant survival rate from baseline to 2 year end of study visit.</li> <li>Knee Society Score 2011</li> <li>Quality of Life (EQ-5D) 5L</li> <li>Forgotten Joint Score (FJS)</li> <li>Hospital Length of Stay</li> <li>Operative Time</li> <li>Radiographic Assessments</li> </ul> |
| Safety Endpoints | The number of occurrences and the frequency of subjects reporting: |
| Length of Study: | Approximately 3 years • 1 year for enrollment and 2 years for follow-up |
| Number of Sites: | Approximately 6 sites |
| Sample Size: Inclusion Criteria: | <ul><li>120 subjects</li><li>1. Subject requires primary total knee arthroplasty with the Journey II BCS</li></ul> |
| | or Cruciate-Retraining (CR) Systems due to degenerative joint disease |



| | | (primary diagnosis of osteoarthritis, post-traumatic arthritis, avascular |
|---|---|---|
| | | necrosis, or rheumatoid arthritis). |
| | 2. | Subject was considered skeletally mature at the time of implantation (at |
| | | least 18 years or older). |
| | 3. | Subject agrees to consent to and to follow the study visit schedule (as |
| | | defined in the study protocol and informed consent form) by signing the |
| | | IRB/EC approved informed consent form. |
| | 4. | Subject plans to be available through two (2) years postoperative follow- |
| | | up. |
| Exclusion Criteria: | 1. | Subject has BMI ≥ 40. |
| | 2. | Subject has condition(s) that may interfere with the TKA survival or |
| | | outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, |
| | | muscular atrophy, uncontrolled diabetes, moderate to severe renal |
| | | insufficiency or neuromuscular disease, or an active, local infection). |
| | 3. | Subject is deemed by investigator to require a constrained or deep dish |
| | | tibial insert. |
| | 4. | Subject has inadequate bone stock to support the device (severe |
| | | osteopenia, history of severe osteoporosis, or severe osteopenia). |
| | 5. | Subject has mental or neurologic condition(s) that may pre-empt the |
| | | ability or willingness to restrict activities. |
| | 6. | Subject is 80 years of age or older. |
| | 7. | Subject is a prisoner or impending incarceration. |



#### BACKGROUND AND STUDY RATIONALE

#### 1.1. Background

Total Knee Arthroplasty (TKA) has become an effective and reliable treatment for arthritis of the knee (1). TKA is associated with low morbidity and mortality, and its effectiveness in reducing joint pain and improving range of motion is well established. In 2014, over 750,000 knee replacements were performed in the US (2).

A significant innovation in TKA has been the introduction of computer navigation and robotic-assisted surgery (3). One such technology is the Navio° Robotic-assisted Surgical System. This system is a semi-autonomous image-free system. During the surgery, the surgeon maps the condylar landmarks and determines alignment indices to define the volume and orientation of bone to be removed. The tools to remove the bone and place the implants are controlled and manipulated by the surgeon with the guidance of a 3-dimensional digital map of the surgical surface.

Originally the Navio° system was launched for use in unicondylar knee replacement only. To date, there have been over 1000 unicondylar knee replacement surgeries using the system. In 2017, Smith & Nephew Inc. expanded the indications for the Navio° system to include TKA. The purpose of this multicenter, prospective study is to evaluate outcomes associated with this new indication.

#### 1.2. Study Rationale

The purpose of this study is to demonstrate superior accuracy with the Navio° Robotic-assisted Surgical System in achieving desired post-operative mechanical alignment, compared to TKA procedures using standard instruments. An additional study purpose is to document clinical and patient-reported outcomes in subjects receiving TKA with the Navio° system.

#### 2. STUDY OBJECTIVES

#### 2.1. Primary Objective

The primary objective of this study is to demonstrate the superiority of the use of the Navio $^{\circ}$  Robotic-assisted Surgical System in the implantation of the JOURNEY $^{\circ}$  II BCS or CR Systems in achieving post-operative mechanical alignment within  $\pm 3^{\circ}$  of target, as compared to TKA procedures using standard instruments.

#### 2.2. Secondary Objectives

Secondary objectives of this study include the generation of safety, performance, and health economic evidence supporting the use of the Navio<sup>o</sup> Robotic-assisted Surgical System in TKA procedures, per the endpoints listed below.

#### 3. STUDY ENDPOINTS

#### 3.1. Primary Endpoint

Post-operative Mechanical Alignment (the proportion of subjects achieving post-operative mechanical alignment, defined as ±3° from target) at the 1 month study visit.



#### 3.2. Secondary Endpoints

The following assessments will be collected at each follow up visit, as described in Section 7.1, Table 1, Schedule of Events.

- Implant survival rate from baseline to 2 year end of study visit.
- Knee Society Score 2011
- Quality of Life (EQ-5D) 5L
- Forgotten Joint Score (FJS)
- Hospital Length of Stay
- Operative Time
- Radiographic Assessments

#### 3.3. Safety Endpoints

The number of occurrences and the frequency of subjects reporting: adverse events (AE), serious adverse events (SAE), adverse device effects (ADE), serious adverse device effects (SADE), unanticipated serious adverse device effects (USADE), and device deficiencies (DevD).

#### 4. STUDY DESIGN

This is a multi-center, prospective cohort study with a comparison to historical control to collect 2-year safety and effectiveness data on 120 subjects, at approximately 6 sites in the United States, who have undergone Navio System-assisted TKA.

Subject data will be evaluated at the pre-operative, operative, one month, six months, one year, and two year follow up visits.

A final analysis will be conducted once all subjects have completed a two year visit.

#### 5. STUDY DEVICE

The Smith & Nephew Navio Robotic-assisted Surgical System aids the surgeon in planning and executing a procedure involving bone preparation for prosthesis implantation. The system is comprised of computer-assisted surgical instrument control, a commercially available surgical drill, image-free navigation, and planning software with standard navigation technology.

The Navio System uses data gathered during the beginning of the surgical procedure (planning phase) to generate a computer model of the knee surface to be remodeled in preparation for the implant. The software uses data collected during the planning phase along with pre-loaded data describing the implant geometry to guide the surgeon in shaping the knee for the selected implant. The Navio system software then allows the surgeon to evaluate the range of motion and fit of the implant prior to finalizing the procedure.

The Navio system software consists of a patient and user management module, a surgical planner, and an intraoperative cutting module. The surgeon uses patient data collected at the surgical site to align the implant and shape the target surface of the bone to accept the intended implant. The Navio system also uses the tracked position of the surgical bur to control its cutting engagement to the bone that is to receive the implant. This cutting control is based on the bur's proximity to the planned target surface of the bone.



The cutting control is achieved in two ways:

- Exposure control adjusts the bur's exposure with respect to a guard. If the surgeon encroaches
  on a portion of bone that is not to be cut, the Navio system retracts the spinning bur behind the
  guard, disabling cutting. The Navio system software also adjusts the depth of the cut by adjusting
  the exposure of the bur outside of the bur guard.
- Speed control regulates the signal transmitted to the drill motor. This limits the speed of the spinning bur or disables bur motion entirely if the target surface has been reached. Bur motion is also disabled if the bur is moved outside of expected cutting boundaries.

The surgeon can alternate between these two cutting control modes. The surgeon can also disable both cutting control modes and operate the Navio system as a standard navigated drill.

The Navio system incorporates a detailed user interface that provides procedure setup, tracking status, visual indicators, and real-time cutting progress during the procedure.

The Navio System is shown below:



| Description | Part Number |
|----------------------------|------------------------------------|
| Tracking Camera and Stand | 110001 |
| Navio System Cart | NPFS-02000, -02010, -02020, -02070 |
| Anspach Drill Foot Control | 120041 |
| Navio System Foot Control | 100460 |
| Navio System Handpiece | 110137 |
| Anspach Drill | 101209 |

The function of each component is as follows:

- Tracking Camera and Stand The mobile infrared tracking camera is used to determine the
  position of the point probe and the surgical bur tip and track their movement by scanning the
  position of reflective trackers relative to the position of trackers mounted on the patient's femur
  and tibia.
- Navio System Cart The mobile cart contains the electronic control system, electrical system integration unit, computer, and uninterruptible power supply (UPS). Navio system carts are



- available in 120 VAC and 220-240 VAC versions. The cart provides storage for the power cord, Anspach drill foot control, and the Navio system foot control. The touchscreen monitor is the primary user interface for the Navio system.
- Anspach Drill Foot Control The Anspach drill foot control is used to control the Anspach drill
  during surgery. The surgeon must press the foot control to activate the bur. The speed of the bur
  is controlled by the Navio system software in speed control mode.
- Navio System Foot Control The Navio system foot control is used as an alternative to the touchscreen monitor when data points are being collected to define landmarks, shape bone, and position the implant prior to surgery.
- Navio System Handpiece The Navio system handpiece controls the position of the Anspach Drill
  and bur relative to the position of the guard and the desired profile of the bone being cut. In
  exposure mode, as the bur nears the target surface of the bone intended to accept the implant,
  the Anspach drill and bur retracts into the guard to prevent further cutting of bone.

The Navio system is intended to assist the surgeon in providing software-defined spatial boundaries for orientation and reference information to anatomical structures during orthopedic procedures. The system is indicated for use in surgical knee procedures, in which the use of stereotactic surgery may be appropriate, and where reference to rigid anatomical bony structures can be determined. These procedures include UKR and patellofemoral arthroplasty. The Navio System is indicated for use with cemented implants only (refer to User Manuals for more detail).

#### 5.1. Surgical Technique

The Navio System is to be used per standard of care at the participating study sites. Each participating investigator will have performed a minimum of 8 Navio TKA procedures prior to enrolling subjects on this study. The Navio System is indicated for Smith & Nephew cemented Total Knee implants, but for the purposed of this study we are restricting the type of implant to the Journey II BCS or Cruciate-Retraining (CR) Systems and compatible S&N patellar implants. The list of acceptable part numbers can be found in Appendix 1. The patella must be resurfaced during the primary TKA procedure.

#### 6. STUDY POPULATION

#### 6.1. Subject Screening & Enrollment

To eliminate the potential for selection bias, Investigators should screen all subjects undergoing a Navio° assisted TKA. In order to do so, only the existing information obtained per standard routine medical procedures will be used. No study-specific screening procedures, activities or questionnaires will be performed during pre-screening.

Once a subject has completed the informed consent procedure and signed the Informed Consent Form, the Principle Investigator (PI), or delegated study research staff, can complete the screening process with the subject. All potential subjects who undergo the screening process will be documented on a Screening and Enrollment Log, on which reasons for exclusion from or denial to participate should be noted. In the event that a subject has a bilateral Navio assisted TKA, only the first knee treated after informed consent will be enrolled in the study.

#### 6.2. Subject Inclusion Criteria

Subjects must meet the following inclusion criteria to be included in the study:



- 1. Subject requires primary total knee arthroplasty with the Journey II BCS or Cruciate-Retraining (CR) Systems due to degenerative joint disease (primary diagnosis of osteoarthritis, post-traumatic arthritis, avascular necrosis, rheumatoid arthritis.
- 2. Subject was considered skeletally mature at the time of cone implantation (at least 18 years or older.)
- 3. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form) by signing the IRB/EC approved informed consent form.
- 4. Subject plans to be available through two (2) years postoperative follow-up.

#### 6.3. Subject Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following exclusion criteria:

- 1. Subject has BMI ≥ 40.
- Subject has condition(s) that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
- 3. Subject is deemed by investigator to require a constrained or deep dish tibial insert.
- 4. Subject has inadequate bone stock to support the device (severe osteopenia, history of severe osteopenia).
- 5. Subject has mental or neurologic condition(s) that may pre-empt the ability or willingness to restrict activities.
- 6. Subject is 80 years of age or older.
- 7. Subject is a prisoner or impending incarceration.



#### 7. STUDY PROCEDURES

#### 7.1. Study Schematic

The intervals and schedule of events are provided in Table 1.

| Schedule of events (*as needed) | Preop | Op/DC | 1 Month | 6 Months | 1 Year | 2 Years |
|---|---|---|---|---|---|---|
| Visit Window | -28<br>days | 0 | 30 <u>+</u> 7<br>days | 182 <u>+</u> 30<br>days | 365 <u>+</u> 60<br>days | 730 <u>+</u> 60<br>days |
| Informed Consent | $\sqrt{}$ | | | | | |
| Inclusion/Exclusion | $\sqrt{}$ | | | | | |
| Demographics/Medical History | $\sqrt{}$ | | | | | |
| Operative Data Collection | | $\sqrt{}$ | | | | |
| Discharge Data Collection | | $\sqrt{}$ | | | | |
| Mechanical Alignment on Long Leg X-<br>rays | $\sqrt{}$ | | $\sqrt{}$ | | | |
| Standard AP, Lateral, and Patellar<br>(Skyline or Merchant) X-rays | | | | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ |
| 2011 Knee Society Score | V | | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ |
| Quality of Life (EQ-5D-5L) | $\sqrt{}$ | | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\checkmark$ |
| Forgotten Joint Score (FJS) | $\sqrt{}$ | | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | $\sqrt{}$ |
| Adverse Event Assessment | | $\sqrt{}$ | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | $\sqrt{}$ |
| End of Study/Exit | | * | * | * | * | * |

<sup>\*</sup> if applicable

#### 7.2. Pre-Operative Visit

Procedures to be completed at the pre-operative visit:

- Confirm informed consent
- Assign a subject study number
- Inclusion/Exclusion
- Demographics and medical history
- 2011 Knee Society Score
- Quality of Life (EQ-5D)
- Forgotten Joint Score
- Perform long leg X-rays to assess Mechanical Alignment

#### 7.3. Surgery

Procedures to be completed at the time of surgery:

- Update information in the Screening and Enrollment Log
- Operative Data including target mechanical alignment
- Discharge Data
- Adverse Event Assessment



#### 7.4. One Month Post-Operative Visit

- Perform long leg X-rays to assess Mechanical Alignment
- 2011 Knee Society Score
- Quality of Life (EQ-5D)
- Forgotten Joint Score
- Obtain and record any AEs occurring from the time of study device implantation
- Adverse Event Assessment

#### 7.5. Six Months, One Year, Two Years Post-Operative

- Perform standard AP, lateral, and patellar X-rays
- 2011 Knee Society Score
- Quality of Life (EQ-5D)
- Forgotten Joint Score
- Obtain and record any AEs occurring from the time of study device implantation
- Adverse Event Assessment
- Collect End of Study Information if applicable

#### 8. SUBJECT COMPLETION AND DISPOSITION

#### 8.1. Screening

Subjects considered potential candidates for the study based on pre-screening will sign an IRB/EC approved Informed Consent Form (ICF) prior to any study activities. The PI, or delegated study research staff, may then complete the first study visit with the subject.

#### 8.2. Enrolled Subject

Subject enrollment occurs at the time of surgery. Every subject that has signed consent, is assigned a Subject ID, and received a total knee implant from the Journey II family with surgical assist from the study device will be considered enrolled in the study.

#### 8.3. Conditions for Study Termination

All reasonable efforts should be made to retain the subjects for the 2 year duration of this study. If the subject has a revision of any component, the subject will be terminated from the study.

#### A. Screening Failure

If a subject has provided consent, completed screening and for any reason is not operated on by the study device and does not receive a total knee implant from the Journey II BCS or Cruciate-Retraining (CR) Systems, the subject will not be considered enrolled in the study.

For these subjects an Inclusion/Exclusion and Informed Consent CRF, Demographics CRF, Medical History CRF, and End of Study CRF need to be completed. However, the CRFs should not be submitted into the Sponsor's database unless the subject signed consent and was assigned a Subject ID.

#### B. Voluntary Withdrawal

Study participation is voluntary and subjects may withdraw at any point during the study without giving their reason for doing so. An End of Study CRF will be completed for all subjects who do not finish the study, and reason for withdrawal will be documented in the form.



#### C. Lost to Follow-Up

Some actively enrolled subjects may not return for follow-up exams due to a variety of reasons. Study personnel must make reasonable efforts to contact the subject and document the following contact attempts prior to declaring a subject to be lost to follow-up: the subject has been contacted according to the site's policies, but no less than 2 documented phone contacts and 1 certified letter without response. Copies of all attempts to reach the subjects per regular mail or email and/or the attempts to contact the subject via other means should be documented and that documentation should be kept with the subjects CRF at the site. A subject will be considered lost to follow-up if he/she does not appear for the scheduled study visit for 2 consecutive visits and study personnel are unable to contact the subject.

#### D. Study Termination by Investigator/Sponsor

The Investigator **may** withdraw subjects from the study for many reasons, including but not limited to the following:

- subject noncompliance to study schematic
- subject lost to follow-up

The Investigator **should** withdraw subjects from the study:

- in case any component of the original Journey II hardware is revised/exchanged
- if the Investigator or the Sponsor stops the study for any reason

For each case, information will be obtained on the End of Study CRF, detailing circumstances leading to the withdrawal.

#### E. Pregnancy

If during the course of the study a subject becomes pregnant, study procedures that are contraindicated during pregnancy and/or lactation (e.g. X-Rays) will not be obtained; however, the subject will continue to be followed for study visits and information will be collected regarding the outcome of the birth.

#### F. Study Site Discontinuation

A specific study site in this multicenter study may also warrant termination under the following conditions:

- non-compliance to Good Clinical Practice (GCP) or protocol
- failure to enroll subjects
- major protocol deviations
- inaccurate or incomplete data
- unsafe or unethical practices
- safety or performance considerations
- investigator involuntarily discontinues participation in study

#### 9. SAFETY REPORTING

Adverse events and device deficiencies, noted by study staff and reported by the subject, and occurring from the time of study device implantation through study completion should be recorded on the appropriate CRFs and reported as below.

#### 9.1. Definitions for safety reporting



#### A. Adverse Event (AE)

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device [1].

This definition includes:

- events related to the investigational medical device or the comparator
- events related to the procedures involved

#### B. Serious Adverse Event (SAE)

A SAE is an adverse event that [1]:

- led to death,
- led to serious deterioration in the health of the subject, that either resulted in:
  - 1) a life-threatening illness or injury, or
  - 2) a permanent impairment of a body structure or a body function, or
  - 3) in-patient or prolonged hospitalization, or
  - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
- led to fetal distress, fetal death or a congenital abnormality or birth defect

Planned hospitalization for a pre-existing condition, or a procedure required by the protocol, without serious deterioration in health, is not considered a serious adverse event.

#### C. Adverse Device Effect (ADE)

An ADE is an adverse event related to the use of an investigational medical device [1].

This definition includes:

- adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.
- any event resulting from use error or from intentional misuse of the investigational medical device.

#### D. Serious Adverse Device Effect (SADE)

An SADE is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event [1].

#### E. Unanticipated Serious Adverse Device Effect (USADE)

A serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report or the clinical investigation plan [1,2].

#### F. Device Deficiency

A device deficiency is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling.

For the purpose of this study, device deficiencies should be reported when they concern any component of the study device or any components of the Journey II implants, as well as its packaging and tools that need to be used during implantation according to the Instructions for Use.



#### G. Revisions

A specially designed Revision Case Report Form will be used in addition to the Adverse Event Form, to document in detail revisions of any of the components of the study device.

#### 9.2. Safety: Investigator's Responsibilities

Investigators shall record adverse events and observed device deficiencies, together with an assessment of seriousness, severity, and relatedness, in the subject's source data. Following, Investigators are responsible for documenting AEs and device deficiencies on the appropriate CRF and submitting them to the Sponsor according to the timelines described here below.

At each contact with the subject, the Investigator must seek information on AEs by specific questioning and, as appropriate, by assessment of the subject. AEs must be recorded in Standard English medical terminology.

Unresolved AEs should be followed by the Investigator until the events are resolved, the subject is lost to follow-up or through to the end of the study, whichever timing occurs first. Unresolved AEs at the end of the subject's participation will be monitored by the Investigator as part of the site's normal standard of care.

The Investigator will categorize AEs as mild, moderate or severe based on the following definitions:

- Mild: the subject is aware of the sign or symptom, but finds it easily tolerated. The event is of
  little concern to the subject and/or little clinical significance. The event is not expected to have
  any effect on the subject's overall health or wellbeing.
- Moderate: the subject has discomfort enough to cause interference with or change in usual activities. The event is of some concern to the subject's health or wellbeing and may require medical intervention and/or close follow-up.
- Severe: the adverse event interferes considerably with the subject's usual activities. The event is of definite concern to the subject and/or poses substantial risk to the subject's health or wellbeing. The event is likely to require medical intervention and/or close follow-up and may be incapacitating or life threatening. Hospitalization and treatment may be required.

The Investigator is responsible for describing the relationship of the AE to Navio (the study device), the implant and the procedure based on the following definitions:

- Unrelated: the event is clearly not related to the study device or procedure
- Possible: the event may or may not be related to the study device or procedure. A relationship cannot be ruled out.
- Definite: the event is clearly related to the study device or procedure.

#### 9.3. Timelines for Submission of Safety Information:

The timelines begin when the Investigator becomes aware of the event.

The Investigator will report to the Sponsor:

- As soon as possible, but no greater than 24 hours upon becoming aware of the event,
   SAEs\*, SADEs, U(S)ADEs and device deficiencies that could have led to a SADE:
  - o if suitable action had not been taken
  - o if intervention had not been made, or
  - if circumstances had been less fortunate



Revisions, within 24 hours upon becoming aware of the event. Sponsor will provide an
explant retrieval kit on becoming aware of a revision and ask the Investigator to return any revised
components for retrieval analysis.

Investigators may also be asked to supply the Sponsor, upon Sponsor's request, with any additional information related to the safety reporting of a particular event.

The Principal Investigator will be responsible for reporting to the IRB/EC of the study site and to the regulatory authorities, SAEs, SADEs and device deficiencies that could have led to a SADE, as required by the national regulations.

#### 9.4. Safety reporting: Sponsor's Responsibilities

Sponsor will provide progress reports on safety events to the Investigator to report to the IRB/EC as required.

In the case of multicenter studies, Sponsor will inform all Investigators in writing of all SAEs that were reported by all sites throughout the clinical investigation and based on perceived risk.

The Sponsor will also, in case of SADEs and device deficiencies that could have led to SADEs, determine whether the risk analysis needs to be updated and assess whether corrective or preventive action is required.

#### 10. STATISTICAL PROCEDURES

#### 10.1. Sample size calculation

Parratte et al. looked at the effects of postoperative mechanical axis alignment on the survival of TKAs. They found that of the 398 TKAs reviewed in the paper there were 292 (73.4%) which post-operatively were defined as mechanically aligned (with a mechanical axis of  $0^{\circ} \pm 3^{\circ}$ ).

This study aims to show superiority in the proportion of TKAs post-operatively defined as mechanically aligned against the reference proportion of 73.4% from above.

It is estimated that the proportion of mechanically aligned TKAs using the Navio system will be around 88%. If this assumption holds then the recruitment of 115 subjects would be sufficient to provide 80% power to show that the lower limit of the two-sided 95% confidence interval for the proportion of mechanically aligned TKAs is greater than 73.4%, hence proving superiority to the reference literature. It is expected that approximately 5% of subjects will be lost to follow up at the 1 month visit and therefore 120 subjects will be recruited for this study.

#### 10.2. General Statistical Considerations

Smith & Nephew's Global Biostatistics group will conduct the statistical analysis for this study and they will prepare Statistical Analysis Plan (SAP). Unless otherwise stated, all significance tests and hypothesis testing will be two-sided, performed at the 5% significance level. Resulting p-values will be quoted and 95% two-sided confidence intervals will be generated where appropriate. All p-values will be rounded to three decimal places, p-values less than 0.001 will be presented as '<0.001' in all tables. Where data summaries are specified, categorical and ordinal variables will be summarized with

frequencies and percentages. Continuous variables will be summarized with the following summary statistics: number of observations, mean, median, standard deviation, minimum and maximum values. All analyses will be performed in SAS 9.4 (or later).



#### 10.3. Missing Data

A complete disposition report, along with the explanation for lost-to-follow-up, death, revision, and withdrawn subjects is to be provided in the Clinical Study Report (CSR). The methods used to handle missing or incomplete data for the efficacy and safety measures will be detailed in the Statistical Analysis Plan (SAP).

#### 10.4. Analysis Populations

All subjects that are operated on by the study device are considered study participants. The following study populations and analysis sets will be defined:

- Safety Population: This population will include all subjects that received the study device and will be used for analysis of demographics, disposition data and safety.
- Modified Intention to Treat Population (mITT): Following the intention to treat principle, this
  population Full Analysis Set (FAS): This will include all subjects that received the study device and
  attended at least one post-baseline assessment. This population will be used for the primary
  analysis of all efficacy endpoints.
- Per Protocol Population (PP): This population will include all subjects that received the study device, meet the inclusion/exclusion criteria, attend all follow-up assessments within the specified window, and have no significant protocol deviations. Subjects that are required to be withdrawn from the study under the protocol (e.g. due to revision) will be included regardless of attendance of follow-up visits unless they are deemed to have significant protocol deviations or failed to meet the inclusion/exclusion criteria. This population will be used as secondary analysis of all efficacy endpoints.

#### 10.5. Analysis of Primary Endpoint

The primary endpoint of the study is the proportion of subjects achieving post-operative mechanical alignment, defined as  $\pm 3^{\circ}$  from target, assessed at the 1 month study visit, and after undergoing a Navio assisted TKA.

The proportion defined above will be presented along with the associated two-sided 95% confidence interval, to be calculated using exact binomial methods.

Superiority of the proportion of subjects achieving post-operative mechanical alignment, after undergoing a Navio assisted TKA against those in the reference literature (Parratte et al.)<sup>7</sup> will be achieved if the lower limit of the two-sided 95% confidence interval is greater than 73.4%.

Mechanical alignment will also be summarized using summary statistics.

#### 10.6. Analysis of Secondary Endpoints:

Implant survival rate will be assessed for a final analysis using the number and proportion of subjects who had no implant revisions by the 2-year time point, the associated 95% confidence intervals will be calculated using exact binomial methods. Time to occurrence of revisions will also be analyzed using Kaplan-Meier survival analysis.

KSS, EQ-5D-5L, and FJS scores will be analyzed separately at the end of study using Repeated Measures ANOVA models, prognostic and baseline factors will be adjusted for.



Length of hospital stay, operative time (both skin to skin time and anesthetic time), and radiographic assessments will be assessed using summary statistics. Trends in operative time measures for individual investigators over the course of the study will be assessed.

#### 10.7. Analysis of Safety Endpoints:

The safety endpoints for this study are the number of occurrences and the frequency of subjects reporting: adverse events (AE), serious adverse events (SAE), adverse device effects (ADE), serious adverse device effects (SADE), unanticipated serious adverse device effects (USADE) and device deficiencies (DevD).

In addition, for each event, the following will be summarised: seriousness, the relationship to the investigational device (Navio), relationship to implant, relationship to study procedure, outcome and either the duration of the resolved events or the duration of the events at study completion.

#### 11. ETHICAL CONSIDERATIONS

#### 11.1. Ethical Approval

In accordance with the Declaration of Helsinki and local regulations of the participating countries, sites must gain written IRB/EC approval prior to enrolling research participants in the study.

#### 11.2. Protocol Amendments

Neither the Investigator nor the Sponsor will modify this protocol without mutual agreement. After agreement to initiate the modification - in the form of a protocol amendment - the Investigator agrees not to implement this modification until instructed to do so by the Sponsor. It will be necessary to obtain IRB/EC approval prior to implementation of any change in the protocol that may affect the scientific soundness or the rights, safety, or welfare of the subjects involved. Notification shall be submitted to the IRB/EC of the study site by the Investigator.

#### 11.3. Informed Consent

All study subjects must sign an IRB/EC approved ICF according to 2011:ISO14155 guidelines, GCP guidelines and all applicable national regulations. Potential subjects must be informed as to the purpose of the study and the potential risks and benefits known or that can be reasonably predicted or expected as described in the written consent form. The subject shall have sufficient opportunity to consider participation in the study; a subject cannot be led to believe that he/she is waiving his/her rights as a subject or the liability of the Sponsor or Investigator. Subjects are then invited to sign and date the consent form, indicating their consent for enrollment. The Investigator will retain the original copy of the signed consent form in the study files. A duplicate copy shall be provided to the subject.

#### 11.4. Risk - Benefit Analysis

#### A. Study Related Risks

#### Possible risks that may occur as a result of study procedures are:

- Subjects will be asked to complete questionnaires; however these are not interventional procedures and are not expected to add significant time to any appointments.
- This study involves the use of x-ray evaluation. X-ray exposure is cumulative over a lifetime and total exposure should be kept to a minimum. However, if the x-ray exposure when participating in the



- study is equivalent to the exposure the subject would receive if they chose not to participate in the study, there is no additional risk associated with this study.
- As a result of participating in the study there could be a risk of loss of protected subject information confidentiality. All applicable confidentiality standards and data protection and privacy laws will be followed by the Sponsor to ensure that data collected is handled in confidence. Data will be coded and handled only by appropriately qualified and authorized personnel.

Risks related to the general surgical procedures are not considered here because these could be present regardless of participation into the study.

#### B. Study Related Benefits

Because the surgery and all the follow-up visits are the same as if the subject would not participate in this study, there are no additional medical benefits associated with participating in this study. The information gained from this study may help improve the treatment of people that need to undergo TKA.

#### 12. MONITORING PROCEDURES

#### 12.1. Source Documentation

Investigators are responsible for obtaining and maintaining complete subject health information in the medical record for each subject (source documents). Examples of source documents follows: hospital records, clinic and office charts, memoranda, dispensing records, subject questionnaires, clinic evaluation transcriptions, operative notes, x-rays, radiology reports, blood collection reports and shipment records, and research subject files.

Original CRFs may be used as source documents only in the case of 2011 Knee Society Score, Quality of Life (EQ-5D) and the Forgotten Joint Score.

The Principal Investigator shall ensure that clinical records are clearly marked to indicate that the subject is enrolled in a particular clinical study and if he/she completed per protocol or discontinued early and the reason.

#### 12.2. Direct Access

This study may be monitored by the Sponsor or a qualified person designated by the Sponsor. This qualified person could be an employee of the Sponsor or of a contract research organization (Sponsor's agent).

The investigator will provide Sponsor, Sponsor's agents, IRB/EC and regulatory agencies with direct access to all source data/documents to permit study-related monitoring, audits, IRB/EC review, and regulatory inspections.

#### 12.3. Site Qualification Visit

A site qualification visit may be performed by the Sponsor prior to the execution of a clinical agreement to ensure that all Investigators have the appropriate training, staff, facilities and resources to adequately conduct the study.

#### 12.4. Site Initiation Visit



A site initiation visit to provide training on the specifics of the study, site obligations and expectations of study conduct will be performed by the Sponsor. No screening or other study procedures may be performed prior to the execution of the Clinical Study Agreement and documented IRB/EC approval.

#### 12.5. Interim Monitoring Visits

The Sponsor or its designee will conduct the appropriate site visits at the appropriate intervals. The clinical investigation will be monitored to ensure that: the rights and wellbeing of the subjects are protected; the reported data are accurate, complete, and verifiable from the source documents; and the study is conducted in compliance with currently approved protocol, with GCP regulations, and with applicable regulatory requirements. Detailed monitoring requirements will be documented within the Clinical Monitoring Plan for this study.

#### 12.6. Closeout Visit

A study close out visit will be performed by the Sponsor or designee to retrieve and account for all remaining clinical data and to resolve outstanding queries. During study close-out, the monitor will review investigator files to ensure required documents and records are on file, confirm the disposition of any other ancillary items used for the study, and review regulatory requirements regarding records retention and IRB/EC reporting requirements.

#### 12.7. Sponsor Audits and Regulatory Inspection

The Sponsor's agents, IRB/EC and regulatory agencies may audit study data. The site must accommodate audit requests, notify the Sponsor of any requests as soon as they are received, and provide direct access to study records during the audit.

#### 12.8. Data Handling and Record Keeping Requirements

Case report forms (CRFs) will be supplied by the Sponsor. Subjects will be identified by a study number and subject identification code. Only the Investigator site will have the key to identify individual subjects. The Investigator is responsible for the timely and accurate completion of CRFs. All documents related to the study must be securely archived at the study site or in a central archive.

Data required according to this protocol are to be recorded on the case report forms (CRFs) at the time of the scheduled visits. Once a subject is enrolled, completed CRFs should be sent to the Sponsor, either by fax or by e-mail, as soon as possible, and is generally expected within 10 working days upon completion of the CRFs.

#### 12.9. Data Recording and Record Retention

Clinical research records shall be stored in a manner that ensures privacy, confidentiality, security and accessibility of the records both during and after the conduct of the study. The Investigator/Institution will take measures to prevent accidental or premature destruction of those documents. The investigator must retain essential study documents for at least 2 years after the latest of the following: the date the study is terminated or completed or the date the documents are no longer needed to support a premarket approval application. If the Investigator needs to dispose of the documents, the Sponsor should be contacted for approval prior to disposal or destruction. For discontinued product, the essential documents will be retained until at least 2 years have elapsed since the formal discontinuation (via notification of the FDA or other regulatory agency) of clinical development of the investigational product. The investigator will retain these documents for a longer period if required by the applicable local laws.



If the responsible investigator retires, relocates, or withdraws from responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

#### 13. DEVIATIONS FROM PROTOCOL

A protocol deviation is an instance of failure, intentionally or unintentionally, to follow the requirements of the protocol. Protocol deviations include but are not limited to deviations from inclusion/exclusion criteria, endpoint variable criteria, study visits outside the window, and GCP guidelines.

#### 13.1. Protocol Deviation Reporting Requirements

Deviations must be reported to the Sponsor through the specially designed Protocol Deviation Log as soon as reasonably possible.

When protocol deviations affect the scientific soundness of the study, or the rights, safety or welfare of the study subjects, the Investigator must also report protocol deviations to the IRB/EC of the study site. It is the responsibility of the PI to inform the IRB/EC of the study site of the incident, per local requirements. The local IRB/EC should be consulted on protocol deviation reporting requirements.

Investigators and all study staff (staff at site and at Sponsor) are responsible for ensuring adherence to study protocol. During the monitoring visits, the Sponsor representative will review all deviations with the Investigator. If a deviation is discovered outside of a monitoring visit, it should be evaluated via phone, email or letter. Appropriate measures to address the occurrence, additional monitoring visits, or audit of the study should be taken, which may include defining and implementing a Corrective and Preventive Action (CAPA).

#### 14. Publication policy

The preparation and submission for publication of manuscripts containing the study results shall be in accordance with a process determined by the Clinical Trial Agreements between the study Sponsor and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to the Health Insurance Portability and Accountability Act of 1996.



Page: 24 of 31

#### **BIBLIOGRAPHY**

List all relevant references here.

- 1. ISO 14155:2011
- 2. 21 CFR 812
- 3. ICH Guideline for Clinical Safety Data Management: Definitions and Standards for Expedited Reporting
- 4. Rand, et al, J Arthroplasty (1991) Sep; 6(3);279-84
- 5. 2015 Hip and Knee Implant Review, www.OrthopedicNetworkNews.com
- 6. Dalton, et al, J. Arthroplasty (2016) 31, 1366-1372
- 7. Parratte S, Pagnano MW, Trousdale RT, Berry DJ. Effect of Postoperative Mechanical Axis Alignment on the Fifteen-Year Survival of Modern, Cemented Total Knee replacements. JBJS 2010:92:2143-9



Page: 25 of 31

## **Appendix 1**JOURNEY II BCS and CR Component Part Numbers

## **JOURNEY II FEMORALS**

| Catalog Item Number | Description |
|---------------------|----------------------------------------------|
| 7402-2111 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 1 |
| 7402-2112 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 2 |
| 7402-2113 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 3 |
| 7402-2114 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 4 |
| 7402-2115 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 5 |
| 7402-2116 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 6 |
| 7402-2117 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 7 |
| 7402-2118 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 8 |
| 7402-2119 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 9 |
| 7402-2110 | JOURNEY II BCS FEMORAL OXINIUM RIGHT SIZE 10 |
| 7402-2121 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 1 |
| 7402-2122 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 2 |
| 7402-2123 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 3 |
| 7402-2124 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 4 |
| 7402-2125 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 5 |
| 7402-2126 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 6 |
| 7402-2127 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 7 |
| 7402-2128 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 8 |
| 7402-2129 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 9 |
| 7402-2120 | JOURNEY II BCS FEMORAL OXINIUM LEFT SIZE 10 |
| 7402-4211 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 1 |
| 7402-4212 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 2 |
| 7402-4213 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 3 |
| 7402-4214 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 4 |
| 7402-4215 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 5 |
| 7402-4216 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 6 |
| 7402-4217 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 7 |
| 7402-4218 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 8 |
| 7402-4219 | JOURNEY II BCS FEMORAL COCR RIGHT SIZE 9 |
| 7402-4921 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 1 |
| 7402-4922 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 2 |
| 7402-4923 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 3 |
| 7402-4924 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 4 |
| 7402-4925 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 5 |
| 7402-4926 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 6 |
| 7402-4927 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 7 |



| JOURNEY II FEMORALS | |
|---------------------|-----------------------------------------|
| 7402-4928 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 8 |
| 7402-4929 | JOURNEY II BCS FEMORAL COCR LEFT SIZE 9 |
| 7402-1151 | JOURNEY II CR FEMORAL OXINIUM RT SZ1 |
| 7402-1152 | JOURNEY II CR FEMORAL OXINIUM RT SZ2 |
| 7402-1153 | JOURNEY II CR FEMORAL OXINIUM RT SZ3 |
| 7402-1154 | JOURNEY II CR FEMORAL OXINIUM RT SZ4 |
| 7402-1155 | JOURNEY II CR FEMORAL OXINIUM RT SZ5 |
| 7402-1156 | JOURNEY II CR FEMORAL OXINIUM RT SZ6 |
| 7402-1157 | Journey II CR Femoral Oxinium RT SZ7 |
| 7402-1158 | JOURNEY II CR FEMORAL OXINIUM RT SZ8 |
| 7402-1159 | JOURNEY II CR FEMORAL OXINIUM RT SZ9 |
| 7402-1150 | Journey II CR Femoral Oxinium RT SZ10 |
| 7402-1161 | JOURNEY II CR FEMORAL OXINIUM LT SZ1 |
| 7402-1162 | JOURNEY II CR FEMORAL OXINIUM LT SZ2 |
| 7402-1163 | JOURNEY II CR FEMORAL OXINIUM LT SZ3 |
| 7402-1164 | JOURNEY II CR FEMORAL OXINIUM LT SZ4 |
| 7402-1165 | JOURNEY II CR FEMORAL OXINIUM LT SZ5 |
| 7402-1166 | JOURNEY II CR FEMORAL OXINIUM LT SZ6 |
| 7402-1167 | JOURNEY II CR FEMORAL OXINIUM LT SZ7 |
| 7402-1168 | JOURNEY II CR FEMORAL OXINIUM LT SZ8 |
| 7402-1169 | JOURNEY II CR FEMORAL OXINIUM LT SZ9 |
| 7402-1170 | JOURNEY II CR FEMORAL OXINIUM LT SZ10 |
| 7402-1251 | JOURNEY II CR FEMORAL COCR RT SZ 1 |
| 7402-1252 | JOURNEY II CR FEMORAL COCR RT SZ 2 |
| 7402-1253 | JOURNEY II CR FEMORAL COCR RT SZ 3 |
| 7402-1254 | JOURNEY II CR FEMORAL COCR RT SZ 4 |
| 7402-1255 | JOURNEY II CR FEMORAL COCR RT SZ 5 |
| 7402-1256 | JOURNEY II CR FEMORAL COCR RT SZ 6 |
| 7402-1257 | JOURNEY II CR FEMORAL COCR RT SZ 7 |
| 7402-1258 | JOURNEY II CR FEMORAL COCR RT SZ 8 |
| 7402-1259 | JOURNEY II CR FEMORAL COCR RT SZ 9 |
| 7402-1261 | JOURNEY II CR FEMORAL COCR LT SZ 1 |
| 7402-1262 | JOURNEY II CR FEMORAL COCR LT SZ 2 |
| 7402-1263 | JOURNEY II CR FEMORAL COCR LT SZ 3 |
| 7402-1264 | JOURNEY II CR FEMORAL COCR LT SZ 4 |
| 7402-1265 | JOURNEY II CR FEMORAL COCR LT SZ 5 |
| 7402-1266 | JOURNEY II CR FEMORAL COCR LT SZ 6 |
| 7402-1267 | JOURNEY II CR FEMORAL COCR LT SZ 7 |
| 7402-1268 | JOURNEY II CR FEMORAL COCR LT SZ 8 |
| 7402-1269 | JOURNEY II CR FEMORAL COCR LT SZ 9 |



## JOURNEY II Tibia baseplates

| Catalog Item Number | Description |
|---------------------|-------------------------------------------------|
| 7402-2211 | JOURNEY Tibial Baseplate Nonporous Right Size 1 |
| 7402-2212 | JOURNEY Tibial Baseplate Nonporous Right Size 2 |
| 7402-2213 | JOURNEY Tibial Baseplate Nonporous Right Size 3 |
| 7402-2214 | JOURNEY Tibial Baseplate Nonporous Right Size 4 |
| 7402-2215 | JOURNEY Tibial Baseplate Nonporous Right Size 5 |
| 7402-2216 | JOURNEY Tibial Baseplate Nonporous Right Size 6 |
| 7402-2217 | JOURNEY Tibial Baseplate Nonporous Right Size 7 |
| 7402-2218 | JOURNEY Tibial Baseplate Nonporous Right Size 8 |
| 7193-3635 | JOURNEY Tibial Baseplate Nonporous Right Size 9 |
| 7402-2221 | JOURNEY Tibial Baseplate Nonporous Left Size 1 |
| 7402-2222 | JOURNEY Tibial Baseplate Nonporous Left Size 2 |
| 7402-2223 | JOURNEY Tibial Baseplate Nonporous Left Size 3 |
| 7402-2224 | JOURNEY Tibial Baseplate Nonporous Left Size 4 |
| 7402-2225 | JOURNEY Tibial Baseplate Nonporous Left Size 5 |
| 7402-2226 | JOURNEY Tibial Baseplate Nonporous Left Size 6 |
| 7402-2227 | JOURNEY Tibial Baseplate Nonporous Left Size 7 |
| 7402-2228 | JOURNEY Tibial Baseplate Nonporous Left Size 8 |
| 7193-3634 | JOURNEY Tibial Baseplate Nonporous Left Size 9 |

| JOURNEY II TKA Inserts | |
|---|---|
| Catalog Item Number | Description |
| 7402-7211 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 9MM |
| 7402-7212 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 10MM |
| 7402-7213 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 11MM |
| 7402-7214 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 12MM |
| 7402-7215 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 13MM |
| 7402-7216 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 15MM |
| 7402-7217 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 18MM |
| 7402-7218 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 RIGHT 21MM |
| 7402-7221 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 9MM |
| 7402-7222 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 10MM |
| 7402-7223 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 11MM |
| 7402-7224 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 12MM |
| 7402-7225 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 13MM |
| 7402-7226 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 15MM |
| 7402-7227 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 18MM |
| 7402-7228 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 1-2 LEFT 21MM |



| JOURNEY II TKA Inserts | |
|---|---|
| 7402-7231 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 9MM |
| 7402-7232 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 10MM |
| 7402-7233 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 11MM |
| 7402-7234 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 12MM |
| 7402-7235 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 13MM |
| 7402-7236 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 15MM |
| 7402-7237 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 18MM |
| 7402-7238 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 RIGHT 21MM |
| 7402-7241 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 9MM |
| 7402-7242 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 10MM |
| 7402-7243 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 11MM |
| 7402-7244 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 12MM |
| 7402-7245 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 13MM |
| 7402-7246 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 15MM |
| 7402-7247 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 18MM |
| 7402-7248 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 3-4 LEFT 21MM |
| 7402-7251 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 9MM |
| 7402-7252 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 10MM |
| 7402-7253 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 11MM |
| 7402-7254 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 12MM |
| 7402-7255 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 13MM |
| 7402-7256 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 15MM |
| 7402-7257 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 18MM |
| 7402-7258 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 RIGHT 21MM |
| 7402-7261 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 9MM |
| 7402-7262 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 10MM |
| 7402-7263 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 11MM |
| 7402-7264 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 12MM |
| 7402-7265 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 13MM |
| 7402-7266 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 15MM |
| 7402-7267 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 18MM |
| 7402-7268 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 5-6 LEFT 21MM |
| 7402-7271 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 9MM |
| 7402-7272 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 10MM |
| 7402-7273 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 11MM |
| 7402-7274 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 12MM |
| 7402-7275 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 13MM |
| 7402-7276 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 15MM |
| 7402-7277 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 18MM |
| 7402-7278 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 RIGHT 21MM |
| 7402-7281 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 9MM |
| 7402-7282 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 10MM |
| 7402-7283 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 11MM |
| 7402-7283 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 11MM |



| | JOURNEY II TKA Inserts |
|-----------|-------------------------------------------------------|
| 7402-7284 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 12MM |
| 7402-7285 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 13MM |
| 7402-7286 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 15MM |
| 7402-7287 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 18MM |
| 7402-7288 | JOURNEY II BCS XLPE ARTICULAR INSERT SZ 7-8 LEFT 21MM |
| 7402-5611 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 9MM |
| 7402-5612 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 10MM |
| 7402-5613 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 11MM |
| 7402-5614 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 12MM |
| 7402-5615 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 13MM |
| 7402-5616 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 15MM |
| 7402-5617 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 RIGHT 18MM |
| 7402-5621 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 9MM |
| 7402-5622 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 10MM |
| 7402-5623 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 11MM |
| 7402-5624 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 12MM |
| 7402-5625 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 13MM |
| 7402-5626 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 15MM |
| 7402-5627 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 1-2 LEFT 18MM |
| 7402-5631 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 9MM |
| 7402-5632 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 10MM |
| 7402-5633 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 11MM |
| 7402-5634 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 12MM |
| 7402-5635 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 13MM |
| 7402-5636 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 15MM |
| 7402-5637 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 RIGHT 18MM |
| 7402-5641 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 9MM |
| 7402-5642 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 10MM |
| 7402-5643 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 11MM |
| 7402-5644 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 12MM |
| 7402-5645 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 13MM |
| 7402-5646 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 15MM |
| 7402-5647 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 3-4 LEFT 18MM |
| 7402-5651 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 9MM |
| 7402-5652 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 10MM |
| 7402-5653 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 11MM |
| 7402-5654 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 12MM |
| 7402-5655 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 13MM |
| 7402-5656 | Journey II Cr XLPE Articular Insert SZ 5-6 Right 15MM |



| | JOURNEY II TKA Inserts |
|-----------|-------------------------------------------------------|
| 7402-5657 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 RIGHT 18MM |
| 7402-5661 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 9MM |
| 7402-5662 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 10MM |
| 7402-5663 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 11MM |
| 7402-5664 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 12MM |
| 7402-5665 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 13MM |
| 7402-5666 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 15MM |
| 7402-5667 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 5-6 LEFT 18MM |
| 7402-5671 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 9MM |
| 7402-5672 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 10MM |
| 7402-5673 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 11MM |
| 7402-5674 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 12MM |
| 7402-5675 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 13MM |
| 7402-5676 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 15MM |
| 7402-5677 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 RIGHT 18MM |
| 7402-5681 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 9MM |
| 7402-5682 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 10MM |
| 7402-5683 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 11MM |
| 7402-5684 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 12MM |
| 7402-5685 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 13MM |
| 7402-5686 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 15MM |
| 7402-5687 | JOURNEY II CR XLPE ARTICULAR INSERT SZ 7-8 LEFT 18MM |

| Patellar Implants | | |
|-----------------------------|-----------|-----------|
| J 2 Patella Resurfacing | | |
| | Catalog # | Size (mm) |
| | 74024826 | 26 |
| | 74024829 | 29 |
| | 74024832 | 32 |
| | 74024835 | 35 |
| | 74024838 | 38 |
| | 74024841 | 41 |
| J 2 Patella, Biconvex | | |
| | 74024623 | 23 |
| | 74024626 | 26 |
| | 74024629 | 29 |
| | 74024632 | 32 |
| Genesis 2 Patella, Biconvex | | |
| | 71420566 | 23 |
| | 71420568 | 26 |
| | 71420570 | 29 |



| Patellar Implants | | |
|--------------------------------|----------|----|
| | 71420572 | 32 |
| Genesis 2 Patella, Resurfacing | | |
| | 71420580 | 26 |
| | 71420574 | 29 |
| | 71420576 | 32 |
| | 71420578 | 35 |
| Genesis 2 Patella, Oval | | |
| Resurfacing | | |
| | 71421029 | 29 |
| | 71421032 | 32 |
| | 71421035 | 35 |
| | 71421038 | 38 |
| | 71421041 | 41 |